CLINICAL TRIAL: NCT04614857
Title: Correlation Between Cardiopulmonary Metabolic Cost and Lower Limb Muscle Activity During Inclined Treadmill Gait in the Elderly
Brief Title: Correlation Between Cardiopulmonary Metabolic Cost and Lower Limb Muscle Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-08-147
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-10

CONDITIONS: Gait
Keywords: Muscle activity; Cardiopulmonary metabolic cost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inclined treadmill gait (Experimental): All subjects underwent measurements of muscle activity and respiratory metabolism energy during treadmill walking at a comfortable speed for 5 minutes and measured by three conditions (#0% inclined treadmill gait, #10% inclined treadmill gait, and #16% inclined treadmill gait)
  Interventions: Other: Inclined treadmill gait

INTERVENTIONS:
Other: Inclined treadmill gait — All subjects underwent measurements of muscle activity and respiratory metabolism energy during treadmill walking at a comfortable speed for 5 minutes and measured by three conditions (#0% inclined treadmill gait, #10% inclined treadmill gait, and #16% inclined treadmill gait)

SUMMARY:
The purpose of this study was to determine the effect of lower extremity muscle activity on the increase of cardiopulmonary metabolic cost during inclined treadmill gait in the elderly.

DETAILED DESCRIPTION:
The purpose of this study was to determine the effect of lower extremity muscle activity on the increase of cardiopulmonary metabolic cost during inclined treadmill gait in the elderly.

Metabolic energy expenditure and muscle activity are measured simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Between 65 and 84 years elderly without neurological effects
* Ability to independent gait at least 16% inclined treadmill
* High levels of physical performance (SPPB > 7)

Exclusion Criteria:

* Severe visual impairment or dizziness that increases the risk of falls
* Serious cardiac conditions (hospitalization for myocardial infarction or heart surgery, history of congestive heart failure, documentedserious and unstable cardiac arrhythmias, hypertrophic cardiomyopathy,severe aortic stenosis, angina or dyspnea at rest or during activities ofdaily living)
* Difficult to understand experimental tasks because of extremely severe cognitive impairment
* Recent acute injuries such as fractures within 6 months, or experience in orthopedic surgery such as artificial joint replacement
* Acute injuries such as fractures within 6 months or orthopedic surgery such as artificial joint replacement

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Change on metabolic energy expenditure | 1 hour
  All subjects underwent measurements respiratory metabolism energy during treadmill walking at a comfortable speed for 5 minutes and measured by three conditions (#0% inclined treadmill gait, #10% inclined treadmill gait, and #16% inclined treadmill gait)

SECONDARY OUTCOMES:
Change on muscle activity | 1 hour
  All subjects underwent measurements of muscle activity during treadmill walking at a comfortable speed for 5 minutes and measured by three conditions (#0% inclined treadmill gait, #10% inclined treadmill gait, and #16% inclined treadmill gait)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Hee Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Lee HJ, Lee SH, Lee J, Chang WH, Ryu GH, Kim YH. Correlation between cardiopulmonary metabolic energy cost and lower-limb muscle activity during inclined treadmill gait in older adults. BMC Geriatr. 2021 Aug 23;21(1):469. doi: 10.1186/s12877-021-02401-9. PMID 34425788